CLINICAL TRIAL: NCT01760291
Title: Continued Access to PREVAIL (CAP2)- WATCHMAN Left Atrial Appendage (LAA) Closure Technology
Brief Title: Continued Access to PREVAIL (CAP2) - WATCHMAN Left Atrial Appendage (LAA) Closure Technology
Acronym: CAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S2278
Record Dates: First submitted 2012-11-06; First posted 2013-01-04 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WATCHMAN (Experimental): WATCHMAN LAA Closure Technology
  Interventions: Device: WATCHMAN LAA Closure Technology

INTERVENTIONS:
Device: WATCHMAN LAA Closure Technology

SUMMARY:
To provide additional information about the safety and efficacy of the WATCHMAN LAA Closure Technology

DETAILED DESCRIPTION:
This Continued Access Protocol is a prospective, non-randomized, multicenter study to allow continued access to the WATCHMAN LAA Closure Technology during the data analysis, reporting and review of the PREVAIL pivotal study Pre-Market Application by FDA.

ELIGIBILITY:
Inclusion Criteria: A subject may be enrolled in the study if all of the following inclusion criteria are met:

1. The subject is 18 years of age or older
2. The subject has documented paroxysmal, persistent, or permanent non- valvular atrial fibrillation (i.e., the subject has not been diagnosed with rheumatic mitral valvular heart disease)
3. The subject is eligible for long-term warfarin therapy
4. The subject has a calculated CHADS2 score of 2 or greater; Subjects with a CHADS2 score of 1 may be included if any of the following apply (according to the ACC/AHA/ESC 2006 Guidelines for the Management of

   Subjects with Atrial Fibrillation subjects requiring warfarin therapy):
   * The subject is a female age 75 or older
   * The subject has a baseline Left Ventricular Ejection Fraction (LVEF) > 30% and < 35%
   * The subject is age 65-74 and has diabetes or coronary artery disease
   * The subject is age 65 or greater and has documented congestive heart failure
5. The subject or legal representative is able to understand and willing to provide written informed consent to participate in the trial
6. The subject is able and willing to return for required follow-up visits and examinations

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. The subject requires long-term warfarin therapy (i.e., even if the device is implanted, the subjects would not be eligible to discontinue warfarin due to other medical conditions requiring chronic warfarin therapy). Additionally, a subject with any of the following is excluded:

   * Thrombosis occurring at a young age (<40 years old)
   * Idiopathic or recurrent venous thromboembolism
   * Thrombosis at an unusual site (i.e., cerebral veins, hepatic veins,renal veins, inferior vena cava, mesenteric veins)
   * Family history of venous thromboembolism or of inherited prothrombotic disorder
   * Recurrence or extension of thrombosis while adequately anticoagulated
2. The subject is contraindicated for warfarin therapy or cannot tolerate long-term warfarin therapy
3. The subject is contraindicated or allergic to aspirin
4. The subject is indicated for antiplatelet therapy other than aspirin (for example, a subject indicated for clopidogrel, prasugrel, ticlopidine or ticagrelor due to DES is excluded from enrollment during the dosing regimen). A subject completing a course of antiplatelet therapy may be enrolled after a 7 day washout period
5. The subject had any interventional or surgical procedure within 30 days prior to enrollment or is planning to have an interventional or surgical procedure in the time between the WATCHMAN device implant and 45-day TEE (e.g., cardioversion, ablation, cataract surgery, dental surgery)
6. The subject had a prior stroke or TIA within the 90 days prior to enrollment
7. The subject has had an MI within 90 days prior to enrollment
8. The subject has a history of atrial septal repair or has an ASD/PFO device
9. The subject has an implanted mechanical valve prosthesis
10. The subject suffers from New York Heart Association Class IV Congestive Heart Failure at the time of enrollment
11. The subject has symptomatic carotid disease (defined as >50% stenosis with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is < 50% stenosis
12. The subject's AF is defined by a single occurrence of AF
13. The subject had a transient case of AF (i.e., secondary to CABG, interventional procedure, etc.)
14. The subject's left atrial appendage is obliterated
15. The subject has undergone heart transplantation
16. The subject is currently treated with antibiotics for an active infection
17. The subject has a resting heart rate > 110 bpm
18. The subject has thrombocytopenia (defined as < 70,000 platelets/mm3) or anemia with hemoglobin concentration of < 10 g/dl (i.e., anemia as determined by the investigator which would require transfusion)
19. The subject is actively enrolled in a concurrent clinical study of an investigational drug or investigational device (study specifics may be reviewed with the sponsor prior to enrollment to confirm a concurrent study will not interfere with the outcomes of this study)
20. The subject participated in any of the following studies: PROTECT AF, CAP Registry, or PREVAIL. If the subject received a subject ID number for a prior WATCHMAN study, the subject may not be enrolled. PROTECT AF control subjects may be considered for participation if they have completed 5 year follow up
21. The subject is pregnant or pregnancy is planned during the course of the investigation
22. The subject has a life expectancy of less than two years
23. The subject is unable to complete follow-up visits for the duration of the study

Echo Exclusion Criteria

A subject is excluded from the study if any of the following echocardiographic exclusion criteria (as assessed via TTE and TEE) are met:

1. The subject has LVEF < 30%
2. The subject has intracardiac thrombus or dense spontaneous echo contrast as visualized by TEE and determined by the echocardiographer within 2 days prior to implant
3. The subject has an existing pericardial effusion > 2mm
4. The subject has a high risk patent foramen ovale (PFO) with an atrial septal aneurysm excursion > 15mm or length > 15mm
5. The subject has a high risk PFO with a large shunt defined as early, within 3 beats or substantial passage of bubbles
6. The subject has significant mitral valve stenosis (i.e., MV <1.5 cm2)
7. The subject has complex atheroma with mobile plaque of the descending aorta or aortic arch
8. The subject has a cardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2012-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saibal Kar, M.D., Principal Investigator — Cedars-Sinai Medical Center; Shephal Doshi, M.D., Principal Investigator — Pacific Heart
Locations (3):
- United States (3):
  - Arizona Heart Rhythm Research Center, Phoenix, Arizona
  - Central Baptist Hospital, Lexington, Kentucky
  - Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dukkipati SR, Holmes DR Jr, Doshi SK, Kar S, Singh SM, Gibson D, Price MJ, Natale A, Mansour M, Sievert H, Houle VM, Allocco DJ, Reddy VY. Impact of Peridevice Leak on 5-Year Outcomes After Left Atrial Appendage Closure. J Am Coll Cardiol. 2022 Aug 2;80(5):469-483. doi: 10.1016/j.jacc.2022.04.062. PMID 35902169

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WATCHMAN
Started | 576
Completed | 340
Not Completed | 236

BASELINE CHARACTERISTICS:
Arm/Group | WATCHMAN
Number analyzed (Participants) | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227
  Male | 349
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 542
  More than one race | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 576

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ischemic Stroke
Description: Primary Endpoint Events by Type for Enrolled Subjects
Time Frame: 5 Year Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | WATCHMAN
Number analyzed (Participants) | 576
Participants | 47

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | WATCHMAN
All-Cause Mortality (participants affected / at risk) | 144/576
Serious Adverse Events (participants affected / at risk) | 84/576
Other Adverse Events (participants affected / at risk) | 16/576
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN (N=576)
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 6 (6)
Anemia Requiring Transfusion (General disorders) | 1 (1)
Anemia Requiring Transfusion (Renal and urinary disorders) | 1 (1)
Anemia Requiring Transfusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arrhythmias (Cardiac disorders) | 1 (1)
Bleeding from Varicose Veins (Vascular disorders) | 1 (1)
Bleeding, Other (Vascular disorders) | 2 (2)
Cardiac Perforation (Cardiac disorders) | 3 (3)
Cranial Bleed (Injury, poisoning and procedural complications) | 4 (4)
Cranial Bleed (Nervous system disorders) | 2 (2)
Death - Non-Cardiovascular (Blood and lymphatic system disorders) | 1 (1)
Death - Non-Cardiovascular (Cardiac disorders) | 11 (11)
Death - Non-Cardiovascular (Gastrointestinal disorders) | 2 (2)
Death - Non-Cardiovascular (General disorders) | 3 (3)
Death - Non-Cardiovascular (Infections and infestations) | 12 (12)
Death - Non-Cardiovascular (Injury, poisoning and procedural complications) | 3 (3)
Death - Non-Cardiovascular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11)
Death - Non-Cardiovascular (Nervous system disorders) | 8 (8)
Death - Non-Cardiovascular (Renal and urinary disorders) | 5 (5)
Death - Non-Cardiovascular (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Death - Non-Cardiovascular (Vascular disorders) | 2 (2)
Death- Cardiovascular/Unexplained (Cardiac disorders) | 37 (37)
Death- Cardiovascular/Unexplained (General disorders) | 12 (12)
Death- Cardiovascular/Unexplained (Infections and infestations) | 1 (1)
Death- Cardiovascular/Unexplained (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Death- Cardiovascular/Unexplained (Nervous system disorders) | 6 (6)
Death- Cardiovascular/Unexplained (Renal and urinary disorders) | 1 (1)
Death- Cardiovascular/Unexplained (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Death- Cardiovascular/Unexplained (Vascular disorders) | 5 (5)
Device Thrombus (thrombus on the atrial facing side of the device) (Vascular disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal Bleeding (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 17 (17)
Gastrointestinal Bleeding (Vascular disorders) | 2 (2)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 5 (6)
Hematuria (Renal and urinary disorders) | 5 (6)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Infection (Renal and urinary disorders) | 1 (1)
Major Bleed Requiring Transfusion (Blood and lymphatic system disorders) | 2 (2)
Major Bleed Requiring Transfusion (Gastrointestinal disorders) | 7 (7)
Major Bleed Requiring Transfusion (Injury, poisoning and procedural complications) | 1 (1)
Major Bleed Requiring Transfusion (Vascular disorders) | 19 (22)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Myocardial Infarction (Vascular disorders) | 2 (2)
Oral Bleeding (Gastrointestinal disorders) | 1 (1)
Oral Bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Non-Study Related) (Blood and lymphatic system disorders) | 1 (1)
Other (Non-Study Related) (Cardiac disorders) | 11 (11)
Other (Non-Study Related) (General disorders) | 1 (1)
Other (Non-Study Related) (Infections and infestations) | 4 (4)
Other (Non-Study Related) (Injury, poisoning and procedural complications) | 1 (1)
Other (Non-Study Related) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Other (Non-Study Related) (Nervous system disorders) | 3 (3)
Other (Non-Study Related) (Renal and urinary disorders) | 4 (4)
Other (Non-Study Related) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Non-Study Related) (Vascular disorders) | 1 (1)
Other (Study Related) (Cardiac disorders) | 1 (1)
Other (Study Related) (General disorders) | 1 (1)
Other (Study Related) (Nervous system disorders) | 2 (2)
Other (Study Related) (Renal and urinary disorders) | 2 (2)
Other (Study Related) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Study Related) (Vascular disorders) | 4 (4)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Pericardial Effusion with Cardiac Tamponade (Cardiac disorders) | 8 (8)
Pseudoaneurysm (Vascular disorders) | 2 (2)
Rectal Bleeding (Gastrointestinal disorders) | 2 (2)
Respiratory Failure (Cardiac disorders) | 2 (2)
Respiratory Failure (Infections and infestations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stroke (Hemorrhagic) (Nervous system disorders) | 2 (2)
Stroke (Ischemic) (Nervous system disorders) | 43 (48)
Subdural Hematoma (Injury, poisoning and procedural complications) | 6 (6)
Subdural Hematoma (Nervous system disorders) | 1 (1)
Subdural Hematoma (Vascular disorders) | 1 (1)
Systemic Embolism (Gastrointestinal disorders) | 1 (1)
Systemic Embolism (Vascular disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 7 (7)
Valvular Damage (Nervous system disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN (N=576)
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 1 (1)
Anemia Requiring Transfusion (Vascular disorders) | 1 (1)
Device Thrombus (thrombus on the atrial facing side of the device) (Vascular disorders) | 16 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 4 (4)
Other (Study Related) (General disorders) | 1 (1)
Other (Study Related) (Product Issues) | 1 (1)
Other (Study Related) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 10 (10)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 3 (3)
Stroke (Ischemic) (Nervous system disorders) | 5 (5)
Stroke (Ischemic) (Vascular disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 3 (3)
Transient Ischemic Attack (TIA) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT01760291/Prot_SAP_000.pdf